CLINICAL TRIAL: NCT02040571
Title: The Impact of the Overnight Closed Loop System on Glycemia, Subsequent Day-time Metabolic Control, Insulin Delivery, Counter Regulatory Hormones, Sleep Quality, Cognition and Satisfaction With Treatment, Compared to Open Loop System (Sensor Augmented Pump Therapy) in Both the Clinical Trial Centre and in the Home Setting in Type 1 Diabetes
Brief Title: The Performance of an Artificial Pancreas at Home in People With Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St Vincent's Hospital Melbourne (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other); Medtronic (Industry)
Responsible Party: Principal Investigator, Amin Sharifi, Doctor, St Vincent's Hospital Melbourne
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: U1111-1151-3297
Record Dates: First submitted 2014-01-15; First posted 2014-01-20 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Closed Loop (Experimental)
  Interventions: Device: Closed Loop
- Open Loop (Active Comparator)
  Interventions: Device: Open Loop

INTERVENTIONS:
Device: Closed Loop — A total of 24 participants with T1 Diabetes with sensor augmented insulin pump therapy (SAPT) experience will be recruited from four tertiary hospitals and will enter an un-masked randomised-control crossover trial, with a run-in period followed by two phases (in-hospital and at-home) in each of two stages (Closed Loop and Open Loop in random order). Closed Loop will be the intervention for this study, and its performance will be assessed compared to Open Loop (control treatment).
  Other Names: Closed Loop Glucose-Sensing Insulin-Delivery System
  Arms: Closed Loop
Device: Open Loop — The performance of closed loop system will be compared to open loop system (Sensor Augmented Pump Therapy). Therefore, the Open Loop system will be the control treatment.
  In stage 1 of study, participants are randomized to either closed loop (CL) or open loop (OL). In stage 2, all participants will be crossed to the opposite study arm.
  Throughout the study, those who randomised to OL will receive exactly the same medical attention as the CL participants.
  Other Names: Sensor Augmented Pump Therapy (SAPT)
  Arms: Open Loop

SUMMARY:
The overall aim of the study is to evaluate the performance of Artificial Pancreas or Closed Loop Glucose-Sensing Insulin-Delivery system in comparison to current best available technology represented by Sensor Augmented Pump Therapy (SAPT) in patients with Type 1 Diabetes.

DETAILED DESCRIPTION:
At present, decisions regarding insulin dosing are made by the patient with intermittent support from their medical team. Even with glucose sensor augmented insulin pump therapy (SAPT), representing the most advanced technology currently available, there are emotional and intellectual demands placed upon the patient with the most well-educated, intelligent and diligent patients often unable to perfectly match insulin delivery with their varying requirements. SAPT does improve glycaemia in comparison with insulin pump therapy alone though a significant proportion of patients will still not meet target HbA1c (<7.0%). A Closed Loop (CL) system whereby a computerised algorithm reviews continuous glucose information to determine a T1D patient's insulin requirements and controls insulin delivery will potentially have a major impact upon acute and chronic complications of diabetes as well as upon their quality of life. Overnight glycaemic control, without the added challenge of meals, physical activity and stress, is a realistic initial application of CL in clinical practice.

This study aims to evaluate insulin pump therapy with an overnight CL system in comparison with current best available technology represented by SAPT in Type 1 Diabetes (T1D) patients, in both hospital and then at home. Outcomes of interest will include metabolic control and performance of the Medtronic CL overnight system compared with SAPT (OL), in both the Clinical Trials Centre (CTC) and in the home setting; the relationship between night-time and day-time metabolic control with CL and OL and nocturnal clinical, hormonal and inflammatory factors that may influence subsequent daytime metabolic control; anti-insulin antibody titres and dissociation constants (Rd) upon CL algorithm performance; sleep quality, cognition, satisfaction with treatment and psychological parameters.

A two phase randomised crossover study design is to be employed with the first phase conducted for a single night in the clinical trials centre and the second phase over 5 days in an ambulatory setting.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged greater than 14 years able to provide informed consent.
* T1 Diabetes for a minimum of 6 months (fasting C-peptide levels less than 50 pmol/L).
* HbA1c less than 8.5%.
* Experience with a continuous glucose sensor with established basal insulin infusion patterns, insulin to carbohydrate ratios, regular use of the insulin bolus calculator, can insert/ change sensor by themselves, can recharge transmitter, and has experience in reading real time continuous glucose monitoring (RT-CGM) data.
* Accurate carbohydrate counting.
* Experience in uploading pump information to web.
* Residing in Melbourne or Perth.
* Willing to comply with the study protocol requirements inclusive of those requirements related to participant safety.

Exclusion Criteria:

* Requiring greater than 150 units of insulin/day.
* Diabetic ketoacidosis (DKA) within the past 4 weeks.
* Hypoglycaemic unawareness (Gold score = 4) while on SAPT
* More than 2 severe hypoglycaemic episodes within the last 12 months
* Pregnant or planning pregnancy within study period.
* Renal impairment (eGFR less than 60ml/min).
* Current or recent (less than 4 weeks) inhaled or oral steroid therapy.
* Dermatological conditions (eg psoriasis) involving the region of glucose sensor/ insulin delivery cannula insertion.
* Subject has physical limitations (eg impaired vision) that would compromise operation of the closed loop system.
* Currently involved in another investigational study.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2014-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Continuous glucose monitoring (CGM) time spent in target glycaemic range (4.0-8.0 mmol/L) overnight (0000h - 0800h) during the ambulatory phase (Phase 2) of the study. | Participants will be monitored overnight during the ambulatory phase (Phase 2) of the study, an expected average of 8 hours each night for 4 nights (Day 1-4 of phase 2).
Continuous glucose monitoring (CGM) time spent in target glycaemic range (4.0-8.0 mmol/L) from 2000h-0800h in clinical trial centre (phase 1 of the study). | Participants will be monitored in clinical trial centre (phase 1 of the study), an expected average of 12 hours.

SECONDARY OUTCOMES:
CGM time and area under the curve (AUC) spent above target range (>8.0 mmol/L). | Participants will be monitored from 2000h-0800h in phase 1 of the study, an expected average of 12 hours.
CGM time and area under the curve (AUC) spent above target range (>8.0 mmol/L). | Participants will be monitored overnight (0000h - 0800h) during the ambulatory phase (Phase 2) of the study, an expected average of 8 hours each night for 4 nights (Day 1-4 of phase 2).
CGM time spent in hypoglycaemic range (<4.0 mmol/L and <3.0 mmol/L) and number of episodes of symptomatic hypoglycaemia (indicated by glucose sensor and confirmed by meter glucose). | Participants will be monitored from 2000h-0800h in phase 1 of the study, an expected average of 12 hours.
CGM time spent in hypoglycaemic range (<4.0 mmol/L and <3.0 mmol/L) and number of episodes of symptomatic hypoglycaemia (indicated by glucose sensor and confirmed by meter glucose). | Participants will be monitored overnight (0000h - 0800h) during the ambulatory phase (Phase 2) of the study, an expected average of 8 hours each night for 4 nights (Day 1-4 of phase 2).
CGM measures of glycaemic variability (standard deviation and margin of error). | Participants will be monitored from 2000h-0800h in phase 1 of the study, an expected average of 12 hours.
CGM measures of glycaemic variability (standard deviation and margin of error). | Participants will be monitored overnight (0000h - 0800h) the ambulatory phase (Phase 2) of the study, an expected average of 8 hours each night for 4 nights (Day 1-4 of phase 2).
Number of episodes of blood ketone-positive hyperglycaemia (blood glucose > 15 mmol/L indicated by glucose sensor and confirmed by meter glucose AND blood ketones greater than or equal to 0.6 mmol/L). | Participants will be monitored from 2000h-0800h in phase 1 of the study, an expected average of 12 hours.
Number of episodes of blood ketone-positive hyperglycaemia (blood glucose > 15 mmol/L indicated by glucose sensor and confirmed by meter glucose AND blood ketones greater than or equal to 0.6 mmol/L). | Participants will be monitored overnight (0000h - 0800h) during the ambulatory phase (Phase 2) of the study, an expected average of 8 hours each night for 4 nights (Day 1-4 of phase 2).
Yellow Springs Instrument (YSI) glucose measurements in target range (4.0-8.0 mmol/L). | Participants will be monitored from 2000h-0800h in phase 1 of the study, an expected average of 12 hours.
YSI glucose measurements in hypoglycaemic range (<4.0 mmol/L and <3.0 mmol/L). | Participants will be monitored from 2000h-0800h phase 1 of the study, an expected average of12 hours.
YSI glycaemic variability (standard deviation). | Participants will be monitored from 2000h-0800h in phase 1 of the study, an expected average of 12 hours.
CGM time in glucose target range (4.0-8.0 mmol/L). | Participants will be monitored in daytime (0800h - 0000h) during the phase 1 of the study, an expected average of 16 hours.
CGM time in glucose target range (4.0-8.0 mmol/L). | Participants will be monitored in daytime (0800h - 0000h during the ambulatory phase (Phase 2) of the study, an expected average of 16 hours each day for 4 days (Day 2-5 of phase 2).
CGM time and area under the curve (AUC) spent above target range (>8.0 mmol/L). | Participants will be monitored in daytime (0800h - 0000h) during the phase 1 of the study, an expected average of 16 hours.
CGM time and area under the curve (AUC) spent above target range (>8.0 mmol/L). | Participants will be monitored in daytime (0800h - 0000h) during the ambulatory phase (Phase 2) of the study, an expected average of 16 hours each day for 4 days (Day 2-5 of phase 2)
CGM time spent in hypoglycaemic range (<4.0 mmol/L and <3.0 mmol/L) and number of episodes of symptomatic hypoglycaemia (indicated by glucose sensor and confirmed by meter glucose). | Participants will be monitored in daytime (0800h - 0000h) during the phase 1 of the study, an expected average of 16 hours.
CGM time spent in hypoglycaemic range (<4.0 mmol/L and <3.0 mmol/L) and number of episodes of symptomatic hypoglycaemia (indicated by glucose sensor and confirmed by meter glucose). | Participants will be monitored in daytime (0800h - 0000h) the ambulatory phase (Phase 2) of the study, an expected average of 16 hours each day for 4 days (Day 2-5 of phase 2)
Number of episodes of blood ketone-positive hyperglycaemia (blood glucose > 15 mmol/L indicated by glucose sensor and confirmed by meter glucose AND blood ketones greater than or equal to 0.6 mmol/L). | Participants will be monitored in daytime (0800h - 0000h) the phase 1 of the study, an expected average of 16 hours.
Number of episodes of blood ketone-positive hyperglycaemia (blood glucose > 15 mmol/L indicated by glucose sensor and confirmed by meter glucose AND blood ketones greater than or equal to 0.6 mmol/L). | Participants will be monitored in daytime (0800h - 0000h) the ambulatory phase (Phase 2) of the study, an expected average of 16 hours each day for 4 days (Day 2-5 of phase 2)
Total insulin delivered (based on pump data) | Participants will be monitored from 2000h-0800h in phase 1 of the study, an expected average of 12 hours.
Total insulin delivered (based on pump data). | Participants will be monitored overnight (0000h - 0800h) during the ambulatory phase (Phase 2) of the study, an expected average of 8 hours each night for 4 nights (Day 1-4 of phase 2).
Rates and number of changes in the rate of insulin infusion (based on pump data). | Participants will be monitored from 2000h-0800h in phase 1 of the study, an expected average of 12 hours.
Rates and number of changes in the rate of insulin infusion (based on pump data). | Participants will be monitored overnight (0000h-0800h) during the ambulatory phase (Phase 2) of the study, an expected average of 8 hours each night for 4 nights (Day 1-4 of phase 2).
Closed loop exits (with root cause identified) based on the monitoring by the investigator in real time from a co-located station. | Participants will be monitored from 2000h-0800h in phase 1 of the study, an expected average of 12 hours.
Closed loop exits (with root cause identified) based on the remote monitoring by the investigator. | Participants will be monitored overnight (0000h-0800h) during the ambulatory phase (Phase 2) of the study, an expected average of 8 hours each night for 4 nights (Day 1-4 of phase 2).
Total basal and total bolus insulin delivered (based on pump data) | Participants will be monitored in daytime (0800h - 0000h) the phase 1 of the study, an expected average of 16 hours.
Total basal and total bolus insulin delivered (based on pump data). | Participants will be monitored in daytime (0800h - 0000h) the ambulatory phase (Phase 2) of the study, an expected average of 16 hours each day for 4 days (Day 2-5 of phase 2)
Urinary cortisol and catecholamines on 12-hour urine collection. | Urine sample will be collected between 2000h-0800h in phase 1 of the study.
Urinary cortisol and catecholamines on 12-hour urine collection. | Urine sample will be collected between 2000h-0800h on Day 1 and Day 2 of the ambulatory phase (phase 2) of the study.
Area under the curve for overnight plasma cortisol, growth hormone, glucagon, adrenaline and noradrenaline (based on hourly blood sample collection). | Blood sample will be collected every hour beween 2000h-0800h in phase 1 of the study.
Plasma metanephrines (based on blood sample collection) | At 2000 P.M on Day 1 and 0800 A.M on Day 2 of phase 1 of the study.
Plasma Cortisol, growth hormone, glucagon, adrenaline , noradrenaline and metanephrines based on blood sample collection. | At 0800 A.M on Day 1 and 0800 A.M on Day 5 of phase 2.
Urinary cortisol and catecholamines on 12-hour urine collection. | Urine sample will be collected between 0800h and 2000h on Day 2 of phase 1 of the study.
Urinary cortisol and catecholamines on 12-hour urine collection. | Urine sample will be collected during between 0800h and 2000h of Day 1 and Day 2 of the ambulatory phase (phase 2) of the study.
Sleep quality includes: total sleep time, sleep onset latency, sleep-efficiency, and wakefulness after sleep onset (WASO), total and average activity counts based on Actigraph data. | Actigraph data will be recorded constantly during Phase 1 of the study, an expected average of 24 hours.
Sleep quality includes: total sleep time, sleep onset latency, sleep-efficiency, and wakefulness after sleep onset (WASO), total and average activity counts based on Actigraph data and the Pittsburgh Sleep Quality Index scores. | Actigraph data will be recorded constantly during the ambulatory phase (phase 2) of the study, an expected average of 5 days. Pittsburg Sleep quality Index tool will be done on day 1 and day 5 of phase 2.
Parameters of Inflammation and Oxidative Stress include: Cell Adhesion Molecules, Myeloperoxidase, Oxidised LDL, hs-CRP (based on blood sample collection) and Urinary isoprostanes. | At 2000 P.M on Day 1 and 0800 A.M on Day 2 of phase 1 of the study.
Parameters of Inflammation and Oxidative Stress include: Cell Adhesion Molecules, Myeloperoxidase, Oxidised LDL, hs-CRP (C reactive Protein) based on blood sample collection, and Urinary isoprostanes. | At 0800 A.M on Day 1 and Day 5 of phase 2.
Diabetes Treatment Satisfaction Questionnaire and Semi-Structured Interviews (Questionnaires will generate total scores for treatment satisfaction, fear of hypoglycaemia, diabetes-related distress and hypoglycemia impaired awareness). | On Day 5 of Phase 2 of the study.
Cognitive Assessment: CogState assessment battery outcome measures will be generated. Each battery test point will record participant response times and accuracy rates for all tasks performed. | Twice daily (AM-test and PM-test sessions) on Day 1, Day 2, Day 3, Day 4, and Day 5 of phase 2 of the study.

CONTACTS AND LOCATIONS:
Overall Officials: David Norman O'neal, Principal Investigator — St Vincent's Hospital Melbourne
Locations (1):
- St Vincent's Hospital Melbourne, Fitzroy, Victoria, Australia